CLINICAL TRIAL: NCT05794061
Title: Advances in Neuropsychological Diagnostics
Acronym: NeuroPsiD
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 25C122
Record Dates: First submitted 2023-02-24; First posted 2023-03-31 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Impairment; Dementia; Psychiatric Disorder
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with brain disorders
  Interventions: Behavioral: Neuropsychological instruments
- Healthy controls: Neurologically Healthy Controls
  Interventions: Behavioral: Neuropsychological instruments

INTERVENTIONS:
Behavioral: Neuropsychological instruments — Cognitive and behavioral tests and questionnaires

SUMMARY:
This project is aimed at advancing neuropsychological diagnostics, enriching and modernizing the panorama of both clinical and forensic psychometric testing. The rapid socio-demographic changes, the developments of neuropsychological semiotics and nosography, as well as the growing applicative specialization of neuropsychological assessment make it necessary to introduce further tools to satisfy the diagnostic requests in clinical contexts and more recently in the forensic field (i.e., tests to be administered remotely; bedside screeners; domain-specific in-depth tests; tools for assessing testamentary capacity).

Specifically, the present study aims to: a) develop, calibrate and evaluate the psychometric properties of I and II level clinical and/or forensic neuropsychological tests evaluating instrumental and non-instrumental functions in a sample of neurologically healthy individuals representative of the Italian population ; b) evaluate the cross-sectional and longitudinal clinical usability of the aforementioned tests in clinical samples (patients with neurological and neuropsychiatric pathologies of different etiology).

ELIGIBILITY:
Inclusion Criteria:

* Clinical populations: clinical diagnosis of either neurological (e.g., vascular and degenerative aetiologies) or psychiatric disorders.
* Healthy controls: not applicable

Exclusion Criteria:

* Clinical populations:

  1. Clinical diagnosis not of interest;
  2. Severe general medical conditions;
  3. Uncorrected vision/hearing deficits.
* Healthy controls:

  1. Presence of brain disorders;
  2. Severe general medical conditions;
  3. Uncorrected vision/hearing deficits.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with brain disorders and normotypical.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Brief Assessment of Social Skills-Dementia (BASS-D) | At baseline (i.e., at the enrollment; all participants); after 1 month (for test-retest analyses in neurologically healthy individuals); after 6, 12, and 18 months in participants with neurodegenerative disorders
  A screening test of social cognition in neurodegeneration
Change from baseline in Picture Interpretation Test (PIT) | At baseline (i.e., at the enrollment; all participants); after 1 month (for test-retest analyses in neurologically healthy individuals); after 6, 12, and 18 months in participants with neurodegenerative disorders
  A test of executive functions
Change from baseline in Verbal Reasoning Test (VRT-A) - Absurdity sub-test | At baseline (i.e., at the enrollment; all participants); after 1 month (for test-retest analyses in neurologically healthy individuals); after 6, 12, and 18 months in participants with neurodegenerative disorders
  A test of verbal reasoning
Change from baseline in Brief Executive Language Screen (BELS) | At baseline (i.e., at the enrollment; all participants); after 1 month (for test-retest analyses in neurologically healthy individuals); after 6, 12, and 18 months in participants with neurodegenerative disorders
  A language test
Change from baseline in Bamberg Dementia Screening Test (BDST) | At baseline (i.e., at the enrollment; all participants); after 1 month (for test-retest analyses in neurologically healthy individuals); after 6, 12, and 18 months in participants with neurodegenerative disorders
  A test of global cognitive efficiency
Change from baseline in Testament Definition Scale (TDS) | At baseline (i.e., at the enrollment; all participants); after 1 month (for test-retest analyses in neurologically healthy individuals); after 6, 12, and 18 months in participants with neurodegenerative disorders
  A scale to assess testament representation
Change from baseline in Testamentary Capacity Assessment Tool (TCAT) | At baseline (i.e., at the enrollment; all participants); after 1 month (for test-retest analyses in neurologically healthy individuals); after 6, 12, and 18 months in participants with neurodegenerative disorders
  A test to assess cognitive functions (i.e., memory, executive functions, social cognition, and numerical abilities) at the base of testamentary capacity
Change from baseline in Telephone Interview for Cognitive Status (TICS) | At baseline (i.e., at the enrollment; all participants); after 1 month (for test-retest analyses in neurologically healthy individuals); after 6, 12, and 18 months in participants with neurodegenerative disorders
  A telephone-based screening test of global cognitive efficiency
Change from baseline in Telephone-based Mini-Mental State Examination (I-TEL-MMSE) | At baseline (i.e., at the enrollment; all participants); after 1 month (for test-retest analyses in neurologically healthy individuals); after 6, 12, and 18 months in participants with neurodegenerative disorders
  A telephone-based screening test of global cognitive efficiency
Change from baseline in Telephone-based Global Examination of Mental State (tele-GEMS) | At baseline (i.e., at the enrollment; all participants); after 1 month (for test-retest analyses in neurologically healthy individuals); after 6, 12, and 18 months in participants with neurodegenerative disorders
  A telephone-based screening test of global cognitive efficiency
Change from baseline in Telephone-based Amyotrophic Lateral Sclerosis Cognitive Behavioural Screen (ALS-CBS™-PhV | At baseline (i.e., at the enrollment; all participants); after 1 month (for test-retest analyses in neurologically healthy individuals); after 6, 12, and 18 months in participants with neurodegenerative disorders
  A telephone-based screening test for cognitive functions in ALS
Change from baseline in Telephone-based Frontal Assessment Battery (t-FAB) | At baseline (i.e., at the enrollment; all participants); after 1 month (for test-retest analyses in neurologically healthy individuals); after 6, 12, and 18 months in participants with neurodegenerative disorders
  A telephone-based screening test of executive functions
Change from baseline in Development of the Bizzare Pictures Test (BPT) | At baseline (i.e., at the enrollment; all participants); after 1 month (for test-retest analyses in neurologically healthy individuals); after 6, 12, and 18 months in participants with neurodegenerative disorders
  A new visual test to assess reasoning abilities
Change from baseline in Development Telephone Language Screener (TLS) | At baseline (i.e., at the enrollment; all participants); after 1 month (for test-retest analyses in neurologically healthy individuals); after 6, 12, and 18 months in participants with neurodegenerative disorders
  A new telephone-based test to asses linguistic functions

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Lombardy, Italy